CLINICAL TRIAL: NCT03654001
Title: Efficacy of Albumin Replacement and Balanced Solution in Patients with Septic Shock (the ALBIOSS-BALANCED Trial): a 2-by-2 Factorial, Investigator-initiated, Open- Label, Multicenter, Randomized, Controlled Trial
Brief Title: ALBumin Italian Outcome Septic Shock-BALANCED Trial (ALBIOSS-BALANCED)
Acronym: ALBIOSS-BAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Istituto Di Ricerche Farmacologiche Mario Negri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: RF-2016-02361583
Record Dates: First submitted 2018-08-03; First posted 2018-08-31 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-01

CONDITIONS: Septic Shock
Keywords: Septic Shock; Albumin; Balanced crystalloids
MeSH Terms: conditions — Shock, Septic | interventions — Albumins; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: 2-by-2 factorial design, open-label, multicenter, randomized, controlled trial, in patients with septic shock, as defined according to clinical criteria. Patients will be randomized in a 1:1:1:1 ratio to one of the 4 groups (Albumin + BAL, Albumin + NS, BAL, NS).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Albumin + Balanced (Experimental): Human Albumin In parallel with fluid administration for volume resuscitation, patients will receive 400 ml of 20% albumin solution both at randomization (D0) and at day 1 (D1). Subsequently, from day 2 (D2) until day 90 (D90) or ICU discharge (whichever comes first), 20% albumin will be administered on a daily basis, to maintain serum albumin concentration equal to or greater than 30 g/L, based upon serum albumin determination.
  Balanced crystalloid solutions
  According to the preference and the standard use of the participating center:
  * Ringer Lactate
  * Ringer Acetate
  * Crystalsol
  Interventions: Biological: Albumin; Other: Balanced
- Albumin + Saline (Experimental): Human Albumin In parallel with fluid administration for volume resuscitation, patients will receive 400 ml of 20% albumin solution both at randomization (D0) and at day 1 (D1). Subsequently, from day 2 (D2) until day 90 (D90) or ICU discharge (whichever comes first), 20% albumin will be administered on a daily basis, to maintain serum albumin concentration equal to or greater than 30 g/L, based upon serum albumin determination.
  Normal Saline Na+ 154 mEq/L, Cl- 154 mEq/L (0.9% NaCl).
  Interventions: Biological: Albumin
- Balanced (Experimental): Balanced crystalloid solutions (Ringer Lactate, Ringer Acetate, Crystalsol)
  Interventions: Other: Balanced
- Saline (No Intervention): Normal Saline Na+ 154 mEq/L, Cl- 154 mEq/L (0.9% NaCl).

INTERVENTIONS:
Biological: Albumin — Human Albumin In parallel with fluid administration for volume resuscitation, patients will receive 400 ml of 20% albumin solution both at randomization (D0) and at day 1 (D1). Subsequently, from day 2 (D2) until day 90 (D90) or ICU discharge (whichever comes first), 20% albumin will be administered on a daily basis, to maintain serum albumin concentration equal to or greater than 30 g/L, based upon serum albumin determination.
  Arms: Albumin + Balanced; Albumin + Saline
Other: Balanced — Balanced crystalloid solutions are traditionally crystalloid solutions containing a relatively low concentration of chloride as compared to 0.9% NaCl containing solutions (Normal Saline).
  Other Names: Ringer Lactate, Ringer Acetate, Crystalsol
  Arms: Albumin + Balanced; Balanced

SUMMARY:
Septic shock is a devastating condition often observed in ICU. It is characterized by pro-inflammatory and immune responses, organ failures, high incidence of AKI and lethality. Fluid resuscitation is pivotal as supportive therapy. At present, there are no effective therapies to improve survival of such clinical condition, often characterized by a mortality as high as 40% during the first 90 days from diagnosis.

This project proposes a large 2-by-2 factorial randomized clinical trial testing the efficacy of albumin and the low- chloride balanced crystalloid solutions (either Ringer Lactate, Ringer Acetate, or Crystalsol - BAL) in septic shock.

The investigators have recently concluded a multicenter, randomized trial, the ALBIOS trial, in which, in a post-hoc analysis, albumin, in addition to crystalloids, reduced 90-day mortality in patients with septic shock, as compared to crystalloids alone (Caironi P et al, 2014). Crystalloids with supra-physiological chloride content may deteriorate renal perfusion, increasing the risk of acute kidney injury (AKI) and mortality.

DETAILED DESCRIPTION:
The project will consist of a 2-by-2 factorial, investigator-initiated, open-label, multicenter, randomized, controlled trial, with PROBE design (Prospective Randomized Open Trial with Blinded Evaluation of Outcomes), in patients with septic shock, as defined according to clinical criteria.

Patients will be randomized in a 1:1:1:1 ratio to one of the 4 study groups (Albumin + BAL, Albumin + NS, BAL, NS).

Both the primary endpoints will include events evaluated objectively: 90-day mortality and incidence of AKI, as assessed by KDIGO criteria (KDIGO Acute Kidney Injury Work Group, 2012).

ELIGIBILITY:
Inclusion Criteria:

Patients with septic shock if they meet the two following criteria:

1. Presence of an infection (known or suspected) in at least one site:

   1. Lung
   2. Abdomen
   3. Urinary tract
   4. Others (blood, skin and soft tissues, central nervous system, bones and joints, cardiac system, reproductive organs).
2. Presence of a severe and acute, sepsis-related cardiovascular failure (as assessed by the SOFA score - see Annex 1), requiring vasopressor to maintain mean arterial pressure >=65 mmHg, despite adequate volume resuscitation a) Cardiovascular SOFA score > 2 (3 or 4) If the patient is unable to provide informed consent, she/he can be included in the trial provided that the requirements of ongoing laws are fulfilled; details on this approach are provided in the protocol, par 11.1 and related Annex 3. The patient will be informed about having been included in a clinical trial, as soon as she/he will regain consciousness.

Exclusion Criteria:

1. Age < 18 years
2. Moribund state
3. Known or suspected adverse reaction to albumin administration
4. Septic shock in patients with traumatic brain injury or a clinically active cerebral lesion (known or suspected)
5. Severe congestive heart failure (NYHA III and IV classes)
6. Clinical situations in which the use of albumin is known or supposed to be clinically beneficial (hepatic cirrhosis with ascites, malabsorption syndrome or protein-losing enteropathy, nephrotic syndrome, burns)
7. More than 24 hours after the onset of septic shock
8. Religious objection to the administration of human blood products
9. Presence of chronic end-stage renal disease
10. Severe hyperkalemia (> 6 mmol/L)
11. Known or suspected pregnancy based on patient information
12. Enrollment in other experimental interventional studies
13. Laboratory confirmation for SARS-CoV-2 infection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1319 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
All-cause 90-day mortality | Up to 90 days
  All-cause death from randomization to 90 days
Combined co-primary endpoint | Up to 90 days
  The composite of all-cause death from randomization to 90 days and new occurrence of acute kidney injury (AKI).

SECONDARY OUTCOMES:
ICU mortality | Up to ICU discharge, a median of 9 days
  All-cause death occurring in Intensive Care Unit (ICU)
In-hospital mortality | Up to hospital discharge, a median of 20 days
  All-cause death occurring during hospital stay
1-year mortality | Up to 1 year
  All-cause death from randomization to 1 year
SOFA score | Up to 90 days or ICU discharge - a median of 9 days - whichever comes first
  Severity and incidence of organ failures, as assessed by the Sequential Organ Failure Assessment (SOFA) score. SOFA score is used to determine the extent of organ function in a patient while in the intensive care unit. The score is based on 6 different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. The scale of each score ranges from 0 (no dysfunction) to 4 (maximal dysfunction). The 6 scores are then added up to provide a global score: the highest the value, the worst the condition of the patient.
Incidence of AKI during ICU stay | Up to 90 days or ICU discharge - a median of 9 days - whichever comes first
  Assessed by the Kidney Disease Improving Global Outcome (KDIGO) criteria as any of the following: (1) increase in serum creatinine >=0.3 mg/dl (26.5 mmol/l) within 48 hours; or (2) increase in SCr to >=1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or (3) urine volume <0.5 ml/kg/h for 6 hours.
RRT | Up to 90 days or ICU discharge - a median of 9 days - whichever comes first
  First use of Renal Replacement Therapy (RRT) during ICU stay
Need for vasopressors | Up to 90 days or ICU discharge - a median of 9 days - whichever comes first
  Duration of the need for vasopressors during ICU stay
Mechanical ventilation | Up to 90 days or ICU discharge - a median of 9 days - whichever comes first
  Duration of mechanical ventilation during ICU stay
Secondary infections in ICU | Up to 90 days or ICU discharge - a median of 9 days - whichever comes first
  Incidence of secondary-acquired infections during ICU stay
Duration of stay in ICU | Up to ICU discharge, a median of 9 days
  Duration expressed as number of days spent in ICU
Duration of stay in hospital | Up to hospital discharge, a median of 20 days
  Duration expressed as number of days spent in hospital
1-year functional and physical disability | Up to 1 year
  Evaluation by specific psyco-functional tests

OTHER OUTCOMES:
Severe metabolic acidosis | Up to 90 days or ICU discharge - a median of 9 days - whichever comes first
  Incidence of severe metabolic acidosis
Severe hyperkalemia | Up to 90 days or ICU discharge - a median of 9 days - whichever comes first
  Incidence of severe hyperkalemia

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Caironi, MD, Principal Investigator — AOU S. Luigi Gonzaga, Orbassano; Giacomo Grasselli, MD, Principal Investigator — Policlinico di Milano Ospedale Maggiore | Fondazione IRCCS Ca' Granda
Locations (37):
- Italy (37):
  - Ospedali Riuniti di Ancona, Ancona, AN
  - AOU Policlinico di Bari, Bari, BA
  - ASST Papa Giovanni XXIII, Bergamo, BG
  - ASST BG Est - Ospedale Bolognini, Seriate, BG
  - AST BG Ovest - PO Treviglio, Treviglio, BG
  - Policlinico Sant'Orsola-Malpighi, Bologna, BO
  - Azienda Ospedaliero - Universitaria di Ferrara - Arcispedale Sant'Anna, Cona, FE
  - Ospedale del Mugello, Borgo San Lorenzo, FI
  - Ospedale San Giuseppe, Empoli, FI
  - AOU Careggi, Florence, FI
  - Ospedale Colline dell'Albegna, Orbetello, GR
  - Presidio Ospedaliero di Desio, Desio, MB
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, MB
  - ASST Nord Milano - Ospedale Bassini, Cinisello Balsamo, MI
  - ASST Ovest Milano, Legnano, MI
  - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan, MI
  - ASST Fatebenefratelli - Sacco P.O. Sacco, Milan, MI
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - IRCCS Policlinico San Donato, San Donato Milanese, MI
  - Azienda Ospedaliero-Universitaria di Modena, Policlinico di Modena, Modena, MO
  - AOU Policlinico Paolo Giaccone, Palermo, PA
  - ISMETT, Palermo, PA
  - AOU Pisana, Pisa, PI
  - As FO Azienda sanitaria Friuli Occidentale, Pordenone, PN
  - Fondazione IRCCS Policlinico San Matteo, Pavia, PV
  - IRCCS ASMN Reggio Emilia, Reggio Emilia, RE
  - Ospedale Infermi di Rimini, Rimini, Rimini
  - Fondazione Policlinico Universitario A. Gemelli, Università Cattolica del Sacro Cuore, Roma, RM
  - Ospedale Santa Chiara, Trento, TN
  - Ospedale Santa Croce, Moncalieri, TO
  - Azienda Ospedaliero - Universitaria S. Luigi Gonzaga, Orbassano, TO
  - AOU Città della Salute e della Scienza di Torino, Torino, TO
  - ASU Giuliano Isontina, Trieste, TS
  - Azienda Sanitaria Universitaria Integrata di Udine, Udine, UD
  - Ospedale di Circolo e Fondazione Macchi, Varese, VA
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona, VR
  - Ospedale SS. Antonio e Biagio e Cesare Arrigo, Alessandria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caironi P, Tognoni G, Masson S, Fumagalli R, Pesenti A, Romero M, Fanizza C, Caspani L, Faenza S, Grasselli G, Iapichino G, Antonelli M, Parrini V, Fiore G, Latini R, Gattinoni L; ALBIOS Study Investigators. Albumin replacement in patients with severe sepsis or septic shock. N Engl J Med. 2014 Apr 10;370(15):1412-21. doi: 10.1056/NEJMoa1305727. Epub 2014 Mar 18. PMID 24635772
- [Background] SAFE Study Investigators; Finfer S, McEvoy S, Bellomo R, McArthur C, Myburgh J, Norton R. Impact of albumin compared to saline on organ function and mortality of patients with severe sepsis. Intensive Care Med. 2011 Jan;37(1):86-96. doi: 10.1007/s00134-010-2039-6. Epub 2010 Oct 6. PMID 20924555
- [Background] Mehlman DJ, Bulkley BH, Wiernik PH. Serum alpha-1-fetoglobulin with gastric and prostatic carcinomas. N Engl J Med. 1971 Nov 4;285(19):1060-1. doi: 10.1056/NEJM197111042851907. No abstract available. PMID 4106199
- [Background] Semler MW, Self WH, Rice TW. Balanced Crystalloids versus Saline in Critically Ill Adults. N Engl J Med. 2018 May 17;378(20):1951. doi: 10.1056/NEJMc1804294. PMID 29768150
- [Background] Angus DC, van der Poll T. Severe sepsis and septic shock. N Engl J Med. 2013 Aug 29;369(9):840-51. doi: 10.1056/NEJMra1208623. No abstract available. PMID 23984731